CLINICAL TRIAL: NCT02431754
Title: A Post-Marketing Clinical Study of LY450190 (Combined With Alpha1 Blocker Treatment)
Brief Title: A Study of Tadalafil (LY450190) in Participants With Lower Urinary Tract Symptoms (LUTS) Suggestive of Benign Prostatic Hyperplasia LUTS (BPH-LUTS).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15734; H6D-JE-LVJK (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil; Adrenergic alpha-1 Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental): 5 milligrams (mg) tadalafil administered once daily orally for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
  Interventions: Drug: Tadalafil; Drug: Alpha1 Blocker
- Placebo (Placebo Comparator): Placebo administered once daily orally for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
  Interventions: Drug: Placebo; Drug: Alpha1 Blocker

INTERVENTIONS:
Drug: Tadalafil — Administered orally
  Other Names: LY450190
  Arms: Tadalafil
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Alpha1 Blocker — Administered orally

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the study drug known as tadalafil in participants with benign prostatic hyperplasia who are being treated with an alpha1 blocker. This study has two treatment periods. Participants will receive tadalafil or placebo in each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Present with benign prostatic hyperplasia (BPH; also referred to as BPH-LUTS), based on the disease diagnostic criteria, at study entry.
* Have been treated with a stable dose of an alpha1 blocker (tamsulosin 0.2 mg once daily or silodosin 4 mg twice daily) for at least 8 weeks prior to screening, and continue the same alpha1 blocker at the same dose for the entire duration of the study.
* Are Japanese men.
* Have prostate volume ≥20 milliliters (mL) estimated by transabdominal or transrectal ultrasound at screening.
* Have BPH-LUTS with a Total International Prostate Symptom Score (IPSS) of ≥12 at screening and baseline.
* Have moderate LUTS with urinary peak flow rate (Qmax) ≥4 to ≤15 mL/second at baseline, while meeting both of the following criteria:

  * Prevoid total bladder volume ≥150 to ≤550 mL as assessed by ultrasound
  * Minimum voided volume ≥125 mL
* Demonstrate ≥80% compliance with alpha1 blocker treatment* during the screening period, documented at baseline

  * *Tamsulosin: (Number of doses taken / Number of days to be treated) × 100
  * Silodosin: (Number of doses taken / Number of days to be treated) × 50

Exclusion Criteria:

* Prostate-specific antigen (PSA) >10.0 nanograms (ng)/mL at screening.
* PSA ≥4.0 to ≤10.0 ng/mL at screening if prostate malignancy has not been ruled out to the satisfaction of a urologist.
* Bladder post-void residual (PVR) ≥150 mL by ultrasound determination at screening.
* History of any of the following pelvic conditions:

  * Pelvic surgery or any other pelvic procedure, including radical prostatectomy, pelvic surgery for removal of malignancy, or bowel resection
  * Pelvic radiotherapy
  * Any pelvic surgical procedure on the urinary tract, including minimally invasive BPH-LUTS therapies and penile implant surgery
  * Lower urinary tract malignancy or trauma
* Lower urinary tract instrumentation (including prostate biopsy) within 30 days of screening.
* History of urinary retention or lower urinary tract (bladder) stones within 6 months of screening.
* History of urethral obstruction due to stricture, valves, sclerosis, or tumor at screening.
* History of any of the following treatments within the indicated duration:

  * Antiandrogens within 11 months before screening
  * Dutasteride within 5 months before screening
  * Finasteride within 2 months before screening
  * Any erectile dysfunction treatment previously or currently
  * Any overactive bladder treatment within 4 weeks before screening
* Have a diagnosis or history of prostate cancer at screening.
* Current or history of malignancy at screening (except for treatment-free and relapse-free for ≥3 years at screening).
* Clinical evidence or history of any of the following bladder conditions:

  * Underactive Bladder
  * Detrusor-sphincter dyssynergia (contraction of the detrusor without sphincter relaxation)
  * Interstitial cystitis
* Clinical evidence of any of the following urinary tract conditions:

  * Active urogenital infection
  * Clinically significant microscopic hematuria as determined by a urologist
* History of significant renal insufficiency meeting either of the following:

  * Receiving renal dialysis
  * Creatinine clearance (CLcr) <30 mL/minute
* Clinical evidence of severe hepatic impairment or Aspartate Transaminase (AST) or Alanine Transaminase (ALT) >3 times the upper limit of normal range.
* History of any of the following cardiac conditions:

  * Current or history of angina requiring treatment with nitrates or nitric oxide donors
  * Current or history of unstable angina
  * Positive cardiac stress test without documented evidence of subsequent, effective cardiac intervention (e.g., coronary angioplasty)
* History of any of the following coronary conditions within 90 days of screening:

  * Myocardial infarction
  * Coronary artery bypass graft surgery
  * Percutaneous coronary intervention (for example, angioplasty or stent placement)
* Any evidence or history of heart failure (New York Heart Association [NYHA] ≥ Class III).
* Currently receiving alpha1 blocker therapy for the treatment of hypertension.
* Current or history of any of the following symptoms:

  * Symptoms associated with orthostasis (e.g., recurrent episodes of dizziness, lightheadedness, loss of consciousness, syncope)
  * Causeless fall within 1 year of screening
* Blood pressure-related findings of any of the following at screening:

  * Systolic blood pressure >160 or <90 millimeters of mercury (mm Hg)
  * Diastolic blood pressure >100 or <50 mm Hg
  * Malignant hypertension
  * Uncontrolled arrhythmia

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maebashi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sagamihara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sakai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takatsuki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil/Placebo: 5 milligrams (mg) tadalafil administered once daily (QD) orally for 8 weeks in one of two treatment periods.
  Placebo administered once daily orally for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
- Placebo/Tadalafil: Placebo administered orally QD for 8 weeks in one of two treatment periods.
  5 mg tadalafil administered orally QD for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
Period: Period 1 (8 Weeks)
Arm/Group | Tadalafil/Placebo | Placebo/Tadalafil
Started | 85 | 86
Received at Least One Dose of Study Drug | 85 | 86
Completed | 79 | 82
Not Completed | 6 | 4
Period: Wash-out Period (4 Weeks)
Arm/Group | Tadalafil/Placebo | Placebo/Tadalafil
Started | 79 | 82
Completed | 75 | 82
Not Completed | 4 | 0
Period: Period 2 (8 Weeks)
Arm/Group | Tadalafil/Placebo | Placebo/Tadalafil
Started | 75 | 82
Completed | 74 | 78
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Tadalafil/Placebo: 5 milligrams (mg) tadalafil administered QD orally for 8 weeks in one of two treatment periods.
  Placebo administered once daily orally for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
- Placebo/Tadalafil: Placebo administered once daily orally for 8 weeks in one of two treatment periods.
  5 mg tadalafil administered once daily (QD) orally for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
- Total: Total of all reporting groups
Arm/Group | Tadalafil/Placebo | Placebo/Tadalafil | Total
Number analyzed (Participants) | 85 | 86 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (6.2) | 62.0 (5.8) | 61.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 85 | 86 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 85 | 86 | 171
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 85 | 86 | 171
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 85 | 86 | 171
Current Smoking Habit [Number; unit: participants]
  Yes | 14 | 20 | 34
  No | 71 | 66 | 137

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Preferring Combination Therapy Over Alpha Blocker Alone on the Treatment Preference Questionnaire (TPQ)
Description: TPQ was used to investigate participant's preference between alpha1 blocker monotherapy and combination therapy with alpha1 blocker plus tadalafil. At the end of Treatment Period 2 (or discontinuation), participants were asked to choose a preferred treatment between the two treatments given in Treatment Period 1 and Treatment Period 2.
Time Frame: Week 20
Population: All randomized participants who received at least one dose of study drug and completed the TPQ.
Measure: Number; unit: percentage of participants
Groups:
- Tadalafil/Placebo: 5 milligrams (mg) tadalafil administered once daily (QD) orally for 8 weeks in one of two treatment periods.
  Placebo administered orally QD for 8 weeks in one of two treatment periods. 0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
- Placebo/Tadalafil: Placebo administered orally QD for 8 weeks in one of two treatment periods. 5 milligrams (mg) tadalafil administered once daily (QD) orally for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
Arm/Group | Tadalafil/Placebo | Placebo/Tadalafil
Number analyzed (Participants) | 75 | 82
percentage of participants
  Prefer therapy tadalafil + a1 blocker: number analyzed (Participants) | 33 | 56
  Prefer therapy tadalafil + a1 blocker | 44.0 | 68.3
  Prefer therapy placebo + a1 blocker: number analyzed (Participants) | 42 | 26
  Prefer therapy placebo + a1 blocker | 56.0 | 31.7
Statistical Analysis 1: Comparison: Tadalafil/Placebo vs Placebo/Tadalafil; Test type: Superiority or Other; p = 0.0937, Normal approximation (Z-test)

2. Secondary Outcome: Change From Baseline on the International Prostate Symptom Score (IPSS) Total Score
Description: IPSS Total Score is the sum of Questions 1 through 7 of the IPSS questionnaire. Each question was scored from 0 (none/no symptoms) to 5 (frequent symptoms) for an IPSS Total Score ranging from 0 to 35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline, Week 8
Population: All randomized participants who received at least one dose of study drug and had a baseline and post baseline IPSS measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tadalafil: 5 milligrams (mg) tadalafil administered once daily (QD) orally for 8 weeks in one of two treatment periods.
  0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
- Placebo: Placebo administered orally QD for 8 weeks in one of two treatment periods. 0.2 mg tamulosin once daily or 4 mg silodosin twice daily.
  Participants will remain on stable dose of alpha1 blocker through both treatment periods.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 157 | 156
units on a scale | -2.5 (5.1) | -1.8 (4.2)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.1485, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.69 to 0.26]

3. Secondary Outcome: Change From Baseline on the IPSS Storage (Irritative) Subscore
Description: IPSS Storage (Irritative) subscore was the sum of Questions 2, 4 and 7 of the IPSS questionnaire. Scores ranged from 0 (no irritative symptoms) to 5 (frequent irritative symptoms), with total subscore of the 3 questions for irritative subscore ranging from 0 to 15. Higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline,Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 157 | 156
units on a scale | -0.6 (2.1) | -0.5 (1.9)

4. Secondary Outcome: Change From Baseline on the IPSS Voiding (Obstructive) Subscore
Description: IPSS voiding (obstructive) subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores ranged from 0 (no obstructive symptoms) to 5 (frequent obstructive symptoms), with total subscore of the 4 questions of the obstructive score ranging from 0 to 20. Higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 157 | 156
units on a scale | -2.0 (3.6) | -1.3 (3.0)

5. Secondary Outcome: Change From Baseline on the IPSS Quality of Life Score (IPSS QoL )
Description: IPSS QoL assess participant response to the following question: "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?". Response options are Delighted (0), Pleased (1); Mostly satisfied (2); mixed about equally satisfied and dissatisfied (3); Mostly dissatisfied (4); Unhappy (5); Terrible (6), with a total ranging from 0 to 6 with higher numerical score representing worse Quality of Life from BPH symptom.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 157 | 156
units on a scale | -0.4 (1.1) | -0.4 (0.9)

6. Secondary Outcome: Percentage of Participants With Global Impression of Improvement (PGI-I)
Description: The PGI I is a participant rated instrument that measures the improvement or worsening of the subject's symptoms based on a 7 point scale. A score of "1" indicates that the subject feels his symptoms are "very much better." A score of "4" indicates that the subjects feels "no change" in his symptoms and a score of "7" indicates that the subject feels his symptoms are "very much worse." The percentage of participants who reported a PGI-I score of 1 to 3 are presented in the table below.
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study drug and had a baseline and post baseline PGI-I measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 167 | 161
percentage of participants | 61.1 | 53.4

7. Secondary Outcome: Percentage of Participants With PGI-I (Drug Attributes Questionnaire) on 8 Symptoms for BPH-Lower Urinary Tract Symptoms Improvement
Description: PGI-I (Drug Attributes Questionnaire [DRAQ]) on 8 Symptoms for BPH-Lower Urinary Tract Symptoms.The DRAQ includes the following urinary symptoms: 1. Difficulty to void; 2. Frequent nighttime voiding; 3. Feeling of incomplete emptying; 4. Frequent daytime voiding; 5. Urinary urgency; 6. Taking a long time to urinate; 7. Need abdominal pressure to void; 8. Dribbling, leakage, and/or accidents. Each urinary symptom in the DRAQ will be evaluated by a participant using the PGI-I (discrete variables with seven categories) at the end of each treatment period, compared with how the symptom was before the participant's began taking medication in this study. The percentage of participants who reported a PGI-I (Drug Attributes Questionnaire) score of 1 to 3 are presented in the table below.
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study drug and had a baseline and post baseline PGI-I (DRAQ) measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 167 | 161
percentage of participants
  Difficulty to void - | 44.9 | 37.9
  Frequent nighttime voiding | 48.5 | 42.9
  Feeling of incomplete emptying | 48.5 | 34.8
  Frequent daytime voiding | 42.5 | 37.9
  Urinary urgency | 37.1 | 31.7
  Taking a long time to urinate | 42.5 | 32.9
  Need abdominal pressure to void | 33.5 | 33.5
  Dribbling, leakage, and/or accidents | 26.9 | 27.3

ADVERSE EVENTS:
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/161
Other Adverse Events (participants affected / at risk) | 47/167 | 39/161
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=167) | Placebo (N=161)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 13 (13) | 13 (13)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 4 (4)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Residual urine volume increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Erection increased (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days